CLINICAL TRIAL: NCT03371888
Title: The Platelet -Rich Plasma in the Therapy of Temporomandibular Disorders
Brief Title: The Platelet-Rich Plasma in the Therapy of Temporomandibular Disorders
Acronym: PRP/TMD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Aleksandra Nitecka-Buchta, DMD, PhD, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Silesian MU PRP
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: PRP; Temporomandibular Disorder; Myalgia; Bruxism
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myalgia; Bruxism

STUDY DESIGN:
Intervention Model Description: An intervention performed in experimental group and control group
Who Masked: Participant, Care Provider
Masking Description: double blinded study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP injections (Experimental): Intramuscular injection of Platelet-Rich Plasma into the masseter and temporalis muscle
  Interventions: Biological: Platelet-Rich Plasma intramuscular injections
- 0,9% NaCl injections (Placebo Comparator): Intramuscular injection of 0,9% NaCl into the masseter and temporalis muscle
  Interventions: Biological: Placebo Comparator: 0,9% NaCl intramuscular injections

INTERVENTIONS:
Biological: Platelet-Rich Plasma intramuscular injections — A platelet-rich plasma intramuscular injections into the trigger points of painful muscles were performed.
  Other Names: PRP intramuscular injections
  Arms: PRP injections
Biological: Placebo Comparator: 0,9% NaCl intramuscular injections — A 0,9% NaCl intramuscular injections into the trigger points of painful muscles were performed.
  Other Names: Saline intramuscular injections
  Arms: 0,9% NaCl injections

SUMMARY:
The Platelet-Rich Plasma intramuscular injections into the masseter and temporalis muscle were performed to reduce painful temporomandibular disorder symptoms,such as myalgia, myofascial pain and myofascial pain with referrals. Patients(n=120) were randomly divided into two groups: experimental(n=60) and control group(n=60). In controls injections with 0,9% NaCl were performed. Pain intensity was measured with NPRS (numeriic pain rating scale, 0= no pain, 11= the worst pain that one can imagine) before(0 day), during(10 day) and after(20 day) the therapy with PRP injections.

DETAILED DESCRIPTION:
Patients(n=120) attending The Department of Temporomandibular Disorders and Orthodontics at the Silesian Medical University Poland, Zabrze were enrolled to the study and randomly divided into one of two groups: experimental and control group. Platelet-Rich Plasma(PRP) was prepared for each patient and an intramuscular injections of 0,5 ml PRP into 6 points at each side were performed in experimental group. A follow-up appointment was made after 10 and 20 days and in each visit an injection of PRP or 0,9% NaCl was performed. Pain intensity was measured in NPRS(numeric pain rating scale) and collected data data were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. presence of local myalgia, myofascial pain and myofascial pain with referral within masseter muscles according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) (II.1.A. 1, 2 and 3)
2. patient's agreement for taking part into the research study

Exclusion Criteria:

1. patients being treated with or addicted to analgesic drugs and/or drugs that affect muscle function
2. presence of contraindications for injection therapy
3. patients being treated by neurologist for neurological disorders and/or neuropathic pain and/or headache
4. patients after traumas to the head and neck region in the previous 2 years
5. edentulous patients
6. patients after radiotherapy
7. presence of severe mental disorders
8. pregnancy or lactation
9. pain of dental origin
10. presence of malignancy
11. drug and/or alcohol addiction
12. patients with needle phobia

Ages: 23 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity reduction in VAS scale,(VAS scale 0-10 points) | 14 days
  Decrease in pain intensity in masseter and temporalis muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Nitecka-Buchta, DMD, Principal Investigator — Medical University of Silesia
Locations (1):
- Department of TMD Silesian Medical University, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wright EF, North SL. Management and treatment of temporomandibular disorders: a clinical perspective. J Man Manip Ther. 2009;17(4):247-54. doi: 10.1179/106698109791352184. PMID 20140156
- [Background] Xie X, Zhang C, Tuan RS. Biology of platelet-rich plasma and its clinical application in cartilage repair. Arthritis Res Ther. 2014 Feb 25;16(1):204. doi: 10.1186/ar4493. PMID 25164150
- [Background] Amable PR, Carias RB, Teixeira MV, da Cruz Pacheco I, Correa do Amaral RJ, Granjeiro JM, Borojevic R. Platelet-rich plasma preparation for regenerative medicine: optimization and quantification of cytokines and growth factors. Stem Cell Res Ther. 2013 Jun 7;4(3):67. doi: 10.1186/scrt218. PMID 23759113
- [Background] Salamanna F, Veronesi F, Maglio M, Della Bella E, Sartori M, Fini M. New and emerging strategies in platelet-rich plasma application in musculoskeletal regenerative procedures: general overview on still open questions and outlook. Biomed Res Int. 2015;2015:846045. doi: 10.1155/2015/846045. Epub 2015 May 5. PMID 26075269
- [Background] Stiles CD. The molecular biology of platelet-derived growth factor. Cell. 1983 Jul;33(3):653-5. doi: 10.1016/0092-8674(83)90008-9. PMID 6307524
- [Background] Pihut M, Ferendiuk E, Szewczyk M, Kasprzyk K, Wieckiewicz M. The efficiency of botulinum toxin type A for the treatment of masseter muscle pain in patients with temporomandibular joint dysfunction and tension-type headache. J Headache Pain. 2016;17:29. doi: 10.1186/s10194-016-0621-1. Epub 2016 Mar 24. PMID 27011213
- [Background] Tsai WC, Yu TY, Chang GJ, Lin LP, Lin MS, Pang JS. Platelet-Rich Plasma Releasate Promotes Regeneration and Decreases Inflammation and Apoptosis of Injured Skeletal Muscle. Am J Sports Med. 2018 Jul;46(8):1980-1986. doi: 10.1177/0363546518771076. Epub 2018 May 17. PMID 29772187
- [Background] Mazzocca AD, McCarthy MB, Chowaniec DM, Cote MP, Romeo AA, Bradley JP, Arciero RA, Beitzel K. Platelet-rich plasma differs according to preparation method and human variability. J Bone Joint Surg Am. 2012 Feb 15;94(4):308-16. doi: 10.2106/JBJS.K.00430. PMID 22336969